CLINICAL TRIAL: NCT05659940
Title: Correlation Between a Novel Subset of Neutrophil and Corneal Neovascularization.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KYPJ226
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-11

CONDITIONS: Corneal Neovascularization; Neutrophils
MeSH Terms: conditions — Corneal Neovascularization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood is collected in EDTA coated tube.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy people: Healthy participants whose age and gender are consistent with CNV patients
- CNV patients: Patients who are diagnosed ocular chemical injury coming to Zhongshan Eye Center, Sun Yat-sen University for medical care

SUMMARY:
The purpose of this study is to determine whether a novel subset of neutrophils is correlated with corneal neovascularization in the patients suffered from ocular chemical injury.

DETAILED DESCRIPTION:
Cornea is an avascular transparent tissue providing refractive power for suitable optical performance. But under the condition of injury or infection, the stable microenvironment of ocular surface has been destroyed. Vessels sprout from the limbus to form corneal neovascularization, becoming an important pathological feature and leading cause of blindness. However, the underlying mechanism particular the inflammation-mediated mechanism remains unclear.

With the advancement of single-cell RNA sequencing (scRNA-seq), the investigation of immune cell transcriptomes has obtained great process . Using this advanced method, we identified different immune cell types in the ocular surface microenvironment in corneal neovascularization mouse model. Particularly, we found a specific subset of neutrophils played important role during the corneal angiogenesis. Using the loss-of-function and gain-of-function experiment, we clarified that this novel subset of neutrophils is the major factor that promoting corneal angiogenesis in mouse model. To further explore the relationship between this subset of neutrophils and angiogenesis in human, we plan to detect whether the neutrophil subset is increased in the circulation of chemical burned corneal neovascularization patients.

The main purpose of this study is to assess whether the novel subset of neutrophils has correlation with chemical burned corneal neovascularization. Approximately 33 patients and 33 age matched healthy controls will be recruited. The clinical characteristics, 4ml peripheral blood and the images of slit lamp photography will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed ocular chemical injury with or without corneal neovascularization.

Exclusion Criteria:

1. Those who are diagnosed ocular diseases except for chemical ocular injury, such as uveitis, retinopathy.
2. Those who are diagnosed allergic disease, autoimmune diseases or hematological diseases, infectious disease, such as eczema, systemic lupus erythematosus (SLE), agranulocytosis and viral hepatitis.
3. Those who took immunosuppressive treatments in the past 3 months.
4. Pregnant or nursing women.
5. Those who have serious heart, lung, liver or kidney diseases.
6. Those who have serious systemic diseases.
7. Those who performed ocular surgery (including cataract surgery) in recent three months.
8. Those who have been enrolled in other interventional clinical studies at the same time.
9. Those who are unable to complete the study according to the investigators' requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients who come to Sun Yat-sen University Zhongshan Ophthalmic Center for medical care and healthy people who are volunteers recruited from society
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes of angiogenic neutrophils ratio | Inclusion (Day1) and 1 week
  Peripheral blood is collected in EDTA coated tubes and the red blood cells are lysed. The cells are firstly blocked and then stained the neutrophil subset markers. Flow cytometric analysis is performed at BD LSRFortessa™ Cell Analyzer and cells are analyzed by FlowJo v10 software.

SECONDARY OUTCOMES:
Corneal Neovascularization Score | Inclusion (Day1) and 1 week
  The neovascularization is scored on a scale of 0-3 as previously reported. 0 = no vessels; 1 = neovessels at the corneal limbus; 2 = neovessels spanning approaching the corneal center; 3 = neovessels spanning the central cornea.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China